CLINICAL TRIAL: NCT02731859
Title: EndoBarrier Register Deutschland
Brief Title: EndoBarrier Register Deutschland-Safety and Efficacy of the Endoscopic Duodenal-Jejunal Bypass Sleeve
Acronym: EBRD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EBRD 001
Record Dates: First submitted 2016-01-27; First posted 2016-04-08 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Obesity; Diabetes Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EndoBarrier: All patients with EndoBarrier treatment
  Interventions: Device: Insertion of EndoBarrier for approximately one year

INTERVENTIONS:
Device: Insertion of EndoBarrier for approximately one year — Insertion of EndoBarrier for approximately one year then explantation and follow-up

SUMMARY:
The purpose of this study ist to determine long-term safety and efficacy in weight reduction and improvement of diabetes mellitus of the temporary, endoscopic duodenal-jejunal bypass-sleeve EndoBarrier® in a national registry.

DETAILED DESCRIPTION:
Long-term data are collected by approximately 30 German centers. An electronic Case-Report-Form (eCRF) was designed to collect relevant pre-specified items by the Clinical Trial Center North (CTC). All German sites that have implanted EndoBarrier® since 2010 were invited to provide patient results. Data-acquisition is projected to a period of 5 years and a maximum of 1000 patients. An extension of data-acquisition is planned.

ELIGIBILITY:
Inclusion Criteria:

* clinical decision for treatment with EndoBarrier
* informed consent for registry participation

Exclusion Criteria:

* Patients not meeting the inclusion criteria
* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with either Obesity and/or Diabetes mellitus who are treated with the EndoBarrier
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of HbA1C | From Implantation to at least 2 years follow up
Reduction of Antidiabetic Medication | From Implantation to at least 2 years follow up
Excess weight loss | From Implantation to at least 2 years follow up
Reduction of BMI | From Implantation to at least 2 years follow up
Weight reduction | From Implantation to at least 2 years follow up

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | From Implantation to at least 2 years follow up
  Adverse events associated to implantation, explantation or insertion of EndoBarrier such as bleeding, liver abscess, abdominal pain, nausea, vomiting, duodenal ulcers, duodenal perforation
Improvement of subjective Arthropathia | From Implantation to at least 2 years follow up
  Qualitative Measurement of improvement of subjective Arthropathia, no scale is used
Smoking Status | From Implantation to at least 2 years follow up
Time of implantation and explantation | From Implantation to at least 2 years follow up
Reduction of fasting glucose | From Implantation to at least 2 years follow up
Reduction of fasting insulin | From Implantation to at least 2 years follow up
Reduction of fasting C-Peptide | From Implantation to at least 2 years follow up
Reduction of systolic blood pressure | From Implantation to at least 2 years follow up
Reduction of diastolic blood pressure | From Implantation to at least 2 years follow up
Reduction of antihypertensive medication | From Implantation to at least 2 years follow up
Reduction of total cholesterol | From Implantation to at least 2 years follow up
Reduction of LDL-cholesterol | From Implantation to at least 2 years follow up
Increase of HDL-cholesterol | From Implantation to at least 2 years follow up
Reduction of fasting triglycerides | From Implantation to at least 2 years follow up
Reduction of antihyperlipidemic medication | From Implantation to at least 2 years follow up
Reduction of 25OHD3 | From Implantation to at least 2 years follow up
Reduction of Calcium | From Implantation to at least 2 years follow up
Reduction of Ferritin | From Implantation to at least 2 years follow up
  Ferritin will be measured
Reduction of Hemoglobin | From Implantation to at least 2 years follow up
Reduction of Vitamin B12 | From Implantation to at least 2 years follow up
Reduction of Albumin | From Implantation to at least 2 years follow up
Reduction of Folic acid | From Implantation to at least 2 years follow up
Reduction of Vitamin B1 | From Implantation to at least 2 years follow up
Reduction of Vitamin B6 | From Implantation to at least 2 years follow up
Reduction of CK | From Implantation to at least 2 years follow up
Reduction of AST | From Implantation to at least 2 years follow up
Reduction of ALT | From Implantation to at least 2 years follow up
Reduction of hsCRP | From Implantation to at least 2 years follow up
Duration of implantation process of the EndoBarrier in minutes | From Implantation to at least 2 years follow up
Duration of ithe explantation process of the EndoBarrier in minutes | From Implantation to at least 2 years follow up
Reduction of waist circumference | From Implantation to at least 2 years follow up
Reduction of daily caloric intake | From Implantation to at least 2 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Jens Aberle, Principal Investigator — University hospital Hamburg, Endokrinology
Locations (11):
- Germany (11):
  - Klinikum Augsburg, Augsburg
  - Evangelisches Krankenhaus Köln-Weyertal, Cologne
  - Donau-Ries Klinik Donauwörth, Donauwörth
  - St. Martinus Krankenhaus Düsseldorf, Düsseldorf
  - Klinikum Forchheim, Forchheim
  - Universitätsklinikum Freiburg- Abt. Innere Medizin II, Freiburg im Breisgau
  - Marienhospital Gelsenkirchen, Gelsenkirchen
  - Universitätsmedizin Göttingen, Göttingen
  - Krankenhaus Emmaus-Niesky, Niesky
  - Elisabeth Klinikum Schmalkalde, Schmalkalden
  - Petrus Krankenhaus Wuppertal, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riedel N, Laubner K, Lautenbach A, Schon G, Schlensak M, Stengel R, Eberl T, Dederichs F, Aberle J, Seufert J. Trends in BMI, Glycemic Control and Obesity-Associated Comorbidities After Explantation of the Duodenal-Jejunal Bypass Liner (DJBL). Obes Surg. 2018 Aug;28(8):2187-2196. doi: 10.1007/s11695-018-3144-9. PMID 29504053